CLINICAL TRIAL: NCT00940875
Title: A Randomized, Open-label Study of the Effect of First Line Treatment With Tarceva in Sequential Combination With Gemcitabine, Compared to Gemcitabine Monotherapy, on Progression-free Survival in Elderly or ECOG PS of 2 Patients With Advanced Non-small Cell Lung Cancer.
Brief Title: A Study of Tarceva (Erlotinib) in Sequential Combination With Gemcitabine as First Line Therapy in Patients With Advanced Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was stopped due to slower than expected recruitment.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML22429
Record Dates: First submitted 2009-07-06; First posted 2009-07-16 (Estimated); Results first posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-04

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Gemcitabine

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: erlotinib [Tarceva]; Drug: gemcitabine
- 2 (Active Comparator)
  Interventions: Drug: gemcitabine

INTERVENTIONS:
Drug: erlotinib [Tarceva] — 150mg po on days 15-28 of each 4 week cycle
  Arms: 1
Drug: gemcitabine — 1250mg/m2/day on days 1 and 8 of each 4 week cycle
  Arms: 1
Drug: gemcitabine — 1000mg/m2/day on days 1, 8 and 15 of each 4 week cycle
  Arms: 2

SUMMARY:
This 2 arm study will compare the efficacy and safety of sequential treatment with Tarceva and gemcitabine, and of gemcitabine monotherapy, as first line treatment of elderly patients, or patients with ECOG performance status of 2, with advanced non-small cell lung cancer.Patients will be randomized to receive either sequential gemcitabine 1250mg/m2/day on days 1 and 8 + Tarceva 150mg po on days 15-28 of each 4 week cycle, or gemcitabine monotherapy 1000mg/m2/day on days 1, 8 and 15 of each 4 week cycle. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=70 years of age or with ECOG PS of 2;
* advanced (stage IIIB or IV)non-small cell lung cancer;
* no prior systemic chemotherapy for advanced NSCLC or prior treatment with HER-axis targeted drugs.

Exclusion Criteria:

* active brain metastasis or spinal cord suppression;
* unstable systemic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- Australia (16):
  - Port Macquarie, New South Wales
  - Randwick, New South Wales
  - Sydney, New South Wales
  - Tweed Heads, New South Wales
  - Wollongong, New South Wales
  - Brisbane, Queensland
  - Greenslopes, Queensland
  - Woolloongabba, Queensland
  - Richmond, South Australia
  - Terrace Gardens, South Australia
  - Hobart, Tasmania
  - Bendigo, Victoria
  - Heidelberg, Victoria
  - Melbourne, Victoria
  - Wodonga, Victoria
  - Fremantle, Western Australia

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine Monotherapy: Participants received gemcitabine, 1000 milligrams per square meter (mg/m^2), intravenously (IV), on Days 1, 8, and 15 of Cycles 1-6 (28-day cycles). Participants consented to post-treatment survival follow-up received no further treatment.
- Gemcitabine (G) Plus (+) Erlotinib (E): Participants received gemcitabine, 1250 mg/m^2, IV, on Days 1 and 8 of Cycles 1-6 (28-day cycles). Participants also received erlotinib, 150 mg tablets, orally (PO), once per day on Days 15-28 of Cycles 1-6 (28-day cycles); and 150 mg tablets, PO, once per day thereafter until disease progression, unacceptable toxicity, withdrawal, or study termination (12 months after randomization of the last participant).
Period: Treatment Phase
Arm/Group | Gemcitabine Monotherapy | Gemcitabine (G) Plus (+) Erlotinib (E)
Started | 31 (Disposition analysis includes 3 participants randomized to G+E but received only gemcitabine) | 23 (3 participants randomized to G+E arm received only gemcitabine and were analyzed in Gemcitabine arm)
Completed | 5 | 4
Not Completed | 26 | 19
Not completed — Adverse Event | 9 | 3
Not completed — Death | 3 | 5
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Disease progression | 9 | 11
Not completed — Physician Decision | 1 | 0
Period: Post-Study Treatment
Arm/Group | Gemcitabine Monotherapy | Gemcitabine (G) Plus (+) Erlotinib (E)
Started | 0 | 4
Completed | 0 | 1
Not Completed | 0 | 3
Not completed — Death | 0 | 1
Not completed — Disease Progression | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) (following an intent-to-treat principle): all randomized participants.
Groups:
- Gemcitabine Monotherapy: Participants received gemcitabine, 1000 mg/m^2, IV, on Days 1, 8, and 15 of Cycles 1-6 (28-day cycles). Participants consented to post-treatment survival follow-up received no further treatment.
- Gemcitabine + Erlotinib: Participants received gemcitabine, 1250 mg/m^2, IV, on Days 1 and 8 of Cycles 1-6 (28-day cycles). Participants also received erlotinib, 150 mg tablets, PO, once per day on Days 15-28 of Cycles 1-6 (28-day cycles); and 150 mg tablets, PO, once per day thereafter until disease progression, unacceptable toxicity, withdrawal, or study termination (12 months after randomization of the last participant).
- Total: Total of all reporting groups
Arm/Group | Gemcitabine Monotherapy | Gemcitabine + Erlotinib | Total
Number analyzed (Participants) | 28 | 26 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.8 (8.72) | 72.8 (7.91) | 73.8 (8.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Progression or Death
Description: Progression-free survival (PFS) was defined as the time from randomization to the date of first documentation of progressive disease (PD), according to Response Evaluation Criteria in Solid Tumors (RECIST) version (V) 1.0, or date of death from any cause. PD was defined for target lesions (TLs) as at least a 20 percent (%) increase in the sum of the longest diameter (SLD), taking as reference the smallest SLD recorded since the start of treatment, and for non-target lesions (NTLs) as unequivocal progression of NTLs. Participants without documented PD were censored at the date of last tumor assessment, the last date recorded in the drug log, or the last date of follow-up the participant was known to be progression free, whichever was last. Participants without a post-Baseline (BL) tumor assessment who were known to be alive were censored at the date of randomization.
Time Frame: BL, Day 22 of Cycles 2, 4, and 6 (28-day cycles), every 2 months thereafter until disease progression, participant withdrawal, or study termination (12 months after randomization of the last participant).
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Gemcitabine Monotherapy | Gemcitabine + Erlotinib
Number analyzed (Participants) | 28 | 26
percentage of participants | 96.4 | 96.2

2. Secondary Outcome: Percentage of Participants Who Achieved Confirmed Complete Response (CR) or Partial Response (PR) According to RECIST V 1.0
Description: As per RECIST V 1.0: for TLs, CR was defined as the disappearance of all TLs, and PR was defined as at least a 30% decrease in the SLD of TLs taking as reference the BL SLD. For NTLs, CR was defined as the disappearance of all NTLs and normalization of tumor marker levels. The 95% confidence interval (CI) for one-sample binomial was determined using the Pearson-Clopper Method.
Time Frame: BL, Day 22 of Cycle 2, 4, and 6 (28-day cycles), every 2 months thereafter until disease progression, participant withdrawal, or study termination (12 months after randomization of the last participant).
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemcitabine Monotherapy | Gemcitabine + Erlotinib
Number analyzed (Participants) | 28 | 26
percentage of participants | 7.1 [0.9 to 23.5] | 3.8 [0.1 to 19.6]
Statistical Analysis 1: Comparison: Gemcitabine Monotherapy vs Gemcitabine + Erlotinib; Test type: Superiority or Other; Difference in Response Rates = -3.30, 95% CI 2-sided [-17.5 to 10.9] — The 95% CI for the difference of 2 rates was estimated using the Hauck-Anderson method

3. Primary Outcome: PFS
Description: The median time, in weeks, between randomization and PFS event. Participants without documented PD were censored at the date of last tumor assessment, the last date recorded in the drug log, or the last date of follow-up the participant was known to be progression free, whichever was last. Participants without a post-BL tumor assessment who were known to be alive were censored at the date of randomization. PFS was estimated by using Kaplan-Meier methodology.
Time Frame: BL, Day 22 of Cycles 2, 4, and 6 (28-day cycles), every 2 months thereafter until disease progression, participant withdrawal, or study termination (up to 2 years)
Population: FAS
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Gemcitabine Monotherapy | Gemcitabine + Erlotinib
Number analyzed (Participants) | 28 | 26
weeks | 8.0 [7 to 21] | 10.3 [7 to 15]
Statistical Analysis 1: Comparison: Gemcitabine Monotherapy vs Gemcitabine + Erlotinib; Difference between treatment groups in PFS; Test type: Superiority or Other; p = 0.4798, Log Rank
Statistical Analysis 2: Comparison: Gemcitabine Monotherapy vs Gemcitabine + Erlotinib; Test type: Superiority or Other; p = 0.4805, Wald Test; Hazard Ratio, log = 1.30, 95% CI 2-sided [0.63 to 2.68] — The hazard ratio was estimated using the Cox regression model and stratified by Eastern Cooperative Oncology Group (ECOG) Performance Status (PS), disease stage, histology, and smoking status

4. Secondary Outcome: Percentage of Participants With Non-Progression at Weeks 8 and 16
Description: Non-progression was defined as CR, PR, or stable disease according to RECIST V 1.0: for TLs, CR was defined as the disappearance of all TLs, PR was defined as at least a 30% decrease in the SLD of TLs taking as reference the BL SLD, and SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest SLD recorded since the start of treatment. For NTLs, CR was defined as the disappearance of all NTLs and normalization of tumor marker levels, and SD was defined as the persistence of 1 or more NTLs and/or maintenance of tumor marker levels above the normal limits. The 95% CI for one-sample binomial was determined using the Pearson-Clopper method.
Time Frame: Weeks 8 and 16
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemcitabine Monotherapy | Gemcitabine + Erlotinib
Number analyzed (Participants) | 28 | 26
percentage of participants
  Week 8 | 50.0 [30.6 to 69.4] | 38.5 [20.2 to 59.4]
  Week 16 | 25.0 [10.7 to 44.9] | 11.5 [2.4 to 30.2]
Statistical Analysis 1: Comparison: Gemcitabine Monotherapy vs Gemcitabine + Erlotinib; Week 8; Test type: Superiority or Other; Difference in Response Rates = -11.54, 95% CI 2-sided [-40.3 to 17.2] — The 95% CI for difference of 2 rates was determined using the Hauck-Anderson method
Statistical Analysis 2: Comparison: Gemcitabine Monotherapy vs Gemcitabine + Erlotinib; Week 16; Test type: Superiority or Other; Difference in Response Rates = -13.46, 95% CI 2-sided [-36.0 to 9.0] — The 95% CI for difference of 2 rates was determined using the Hauck-Anderson method

5. Secondary Outcome: Percentage of Participants Who Died
Time Frame: BL, Days 1, 8, and 15 of Cycles 1-6 (28-day cycles), every 28 days thereafter until death, participant withdrawal, or study termination up to 2 years.
Population: FAS
Measure: Number; unit: percentage of participants
Groups:
- Gemcitabine+ Erlotinib: Participants received gemcitabine, 1250 mg/m^2, IV, on Days 1 and 8 of Cycles 1-6 (28-day cycles). Participants also received erlotinib, 150 mg tablets, PO, once per day on Days 15-28 of Cycles 1-6 (28-day cycles); and 150 mg tablets, PO, once per day thereafter until disease progression, unacceptable toxicity, withdrawal, or study termination (12 months after randomization of the last participant).
Arm/Group | Gemcitabine Monotherapy | Gemcitabine+ Erlotinib
Number analyzed (Participants) | 28 | 26
percentage of participants | 92.9 | 76.9

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the median time, in weeks, between randomization and death due to any cause. Participants without documented death were censored at the last date recorded in the drug log, or the last date of follow-up the participant was known to be alive, whichever was last. Participants without a post-BL assessment who were known to be alive were censored at the date of randomization. OS was estimated using Kaplan-Meier methodology.
Time Frame: as for outcome 5
Population: FAS
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Gemcitabine Monotherapy | Gemcitabine + Erlotinib
Number analyzed (Participants) | 28 | 26
weeks | 21.3 [13 to 40] | 17.1 [11 to 37]
Statistical Analysis 1: Comparison: Gemcitabine Monotherapy vs Gemcitabine + Erlotinib; Difference between treatment groups in OS; Test type: Superiority or Other; p = 0.5393, Log Rank
Statistical Analysis 2: Comparison: Gemcitabine Monotherapy vs Gemcitabine + Erlotinib; Test type: Superiority or Other; p = 0.5399, Wald Test; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.38 to 1.66] — The hazard ratio was estimated using the Cox regression model and stratified by ECOG PS, disease stage, histology, and smoking status

7. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time between the first documentation of CR or PR (whichever status was recorded first as assessed by the RECIST V 1.0) until the date of documented disease progression or death. Participants with no documented disease progression or death after confirmed CR or PR were censored at the date of the last tumor assessment or last date of follow-up when the participant was known to be progression free, whichever was last.
Time Frame: as for outcome 5
Population: Data could not be summarized to be included in the data table because there are too few events to calculate a median and confidence intervals.
Arm/Group | Gemcitabine Monotherapy | Gemcitabine+ Erlotinib
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from BL until 28 days after the last date study treatment was received.
Description: All participants who received at least 1 dose/infusion of study treatment and had at least 1 safety assessment performed after BL were included in the safety analysis.
Arm/Group | Gemcitabine Monotherapy | Gemcitabine + Erlotinib
Serious Adverse Events (participants affected / at risk) | 20/31 | 14/23
Other Adverse Events (participants affected / at risk) | 28/31 | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine Monotherapy (N=31) | Gemcitabine + Erlotinib (N=23)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmomary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Pyrexia (General disorders) | 4 | 2
Malaise (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Sudden death (General disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Embolism venous (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Peripheral embolism (Vascular disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine Monotherapy (N=31) | Gemcitabine + Erlotinib (N=23)
Nausea (Gastrointestinal disorders) | 13 | 13
Diarrhoea (Gastrointestinal disorders) | 3 | 12
Constipation (Gastrointestinal disorders) | 6 | 7
Vomiting (Gastrointestinal disorders) | 5 | 6
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Mouth ulceration (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 7 | 10
Oedema peripheral (General disorders) | 8 | 4
Chest pain (General disorders) | 5 | 5
Pyrexia (General disorders) | 3 | 1
Mucosal inflammation (General disorders) | 4 | 3
Pain (General disorders) | 2 | 1
Ill-defined disorder (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Injection site reaction (General disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hilum mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 2
Oral candidiasis (Infections and infestations) | 4 | 1
Cellulitis (Infections and infestations) | 3 | 0
Lung infection (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 15
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 1
Dizziness (Nervous system disorders) | 4 | 2
Headache (Nervous system disorders) | 3 | 2
Lethargy (Nervous system disorders) | 3 | 1
Ataxia (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness postural (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Intention tremor (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 0 | 1
Pyramidal tract syndrome (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Tardive dyskinesia (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 5
Hypertension (Vascular disorders) | 1 | 1
Ischaemic limb pain (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
Blepharitis (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Exophthalmos (Eye disorders) | 0 | 1
Eye irritation (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 1
Foreign body sensation in eyes (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 2
Renal impairment (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Weight decreased (Investigations) | 3 | 2
Alanine aminotransferase increased (Investigations) | 2 | 1
Haemoglobin decreased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Eastern cooperative oncology group performance status worsened (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Platelet count increased (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 6 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 2
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 1 | 3
Anxiety (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 2 | 1
Agitation (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Due to slower than expected recruitment, this study was stopped after 54 patients had been enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.